CLINICAL TRIAL: NCT04083482
Title: Removal of mtDNA in Plasma by Continous Venovenous Hemofiltration in Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Xingui Dai, Critical Care Medicine, First People's Hospital of Chenzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WYJ2019
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Intensive Care Unit
Keywords: Mitochondrial DNA; Sepsis; Continous venovenous hemofiltation; Intensive Care Unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Septic patients require CVVH (Experimental): continuous venovenous hemofiltration. Continuous renal replacement therapy（CRRT）has become routine for patients with chronic renal failure ，AKI，fliud overload as well as oliguria in ICU .Continuous venovenous hemofiltration（CVVH）is the method of chioce for CRRT in critical ill .CVVH has significant beneficial effects on removing inflammatory cytokines ，improving oxygen index ，decreasing vasopressor requirements，increasing cardiac index and regulating immune dysfunction .
  Interventions: Procedure: continous venovenous hemofiltraion

INTERVENTIONS:
Procedure: continous venovenous hemofiltraion — CVVH

SUMMARY:
The plasma level of mtDNA in sepsis is affected by continous venovenous hemofiltation（CVVH）

DETAILED DESCRIPTION:
Continous renal replacement therapy （CRRT）has become routine for patients with chronic renal failure ，AKI，fliud overload as well as oliguria in ICU .In clinical patients ，continous venovenous hemofoiltration （CVVH）is actually the method of chioce for CRRT in critically ill and hemodynamic instable patients .CVVH has significant beneficial effects on removing inflammatory cytokines ，improving oxygen index，increasing cardiac index and regulating immune dysfuntion .

ELIGIBILITY:
Inclusion Criteria:

Adult septic patients undergoing CRRT

Exclusion Criteria:

1. Missing vists
2. transplatation
3. cancer
4. aquired immunodeficiency syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of mtDNA concentration in plasma | befor,6hours, 12hours, after CVVH treatment
  The specimens in the prefilter and postfilter blood as well as in the ultrafiltrate were obtained at the beginning of CRRT (T0) and 6 h (T6h), 12 h (T12h) after the setup of CVVH.

CONTACTS AND LOCATIONS:
Overall Officials: dixian luo, MS, Study Director — Chenzhou First people Hospital
Locations (1):
- The First Hospital of Chenzhou, Chenzhou, Hunan, China